CLINICAL TRIAL: NCT04801745
Title: Effects of a Healthy Vegan Diet Vs. Low Purine Diet, with or Without Amla Fruits (Emblica Officinalis) on Hyperuricemia and Other Cardiometabolic Risk Factors: a Randomized Two-by-two Factorial Trial
Brief Title: Vegan Diet, Amla Fruits and Uric Acid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Tina Hsueh-Ting Chiu, Assistant Professor, Fu Jen Catholic University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2021-02-28; First posted 2021-03-17 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Hyperuricemia; Diet, Healthy; Cardiometabolic Syndrome
Keywords: Vegan diet; Uric acid; Cardiometabolic risk factors; Amla fruits
MeSH Terms: conditions — Hyperuricemia; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Healthy Vegan Diet (Experimental): Education on healthy vegan diet
  Interventions: Other: Healthy vegan diet
- Healthy Vegan Diet with Amla fruits (Experimental): Education on healthy vegan diet, 3g of powdered amla fruits per day
  Interventions: Other: Healthy vegan diet; Other: Amla fruits
- My Plate - Low Purine (Active Comparator): Education on "My Plate" diet with emphasis on choosing low purine protein options.
  Interventions: Other: My Plate - Low Purine
- My Plate - Low Purine with Amla Fruits. (Experimental): Education on "My Plate" diet with emphasis on choosing low purine protein options and with an addition of 3g of amla powder per day.
  Interventions: Other: My Plate - Low Purine; Other: Amla fruits

INTERVENTIONS:
Other: Healthy vegan diet — Participants will attend group lessons and individual nutrition counseling to help them adopt a healthy vegan diet.
  Arms: Healthy Vegan Diet; Healthy Vegan Diet with Amla fruits
Other: My Plate - Low Purine — Participants will attend group lessons and individual nutrition counseling to help them adopt a balanced diet in accordance with my plate, and emphasis on choosing low purine options from the protein food groups.
  Arms: My Plate - Low Purine; My Plate - Low Purine with Amla Fruits.
Other: Amla fruits — Participants will be provided with powdered amla fruits, and will be instructed to take 3g per day.
  Arms: Healthy Vegan Diet with Amla fruits; My Plate - Low Purine with Amla Fruits.

SUMMARY:
This is an intervention study aiming to test the effectiveness of a vegan diet, My Plate with low purine choices, and amla fruits on uric acid and other cardiometabolic risk factors in individuals with high serum uric acid levels.

DETAILED DESCRIPTION:
Ninety-two participants with hyperuricemia will be randomly assigned to one of these 4 diet interventions: (1) vegan, (2) vegan with amla fruits, (3) my plate-low purine, (4) my plate-low purine with amla fruits. During the 3 months intervention phase, participants will attend group lessons and individual nutrition counseling sessions to assist adherence to the diet. At baseline, end of 3 months, and 1 year, participants will be measured on uric acid and other cardiometabolic risk factors, and some nutritional markers. Amla fruits powder, and some foods encouraged in each dietary arm will be provided to enhance adherence during the 3 months intervention phase.

ELIGIBILITY:
Inclusion Criteria:

* Men with serum uric acid > 7mg/dL
* Women with serum uric acid > 6mg/dL
* Willing to make diet changes according to dietary interventions

Exclusion Criteria:

* Age <19
* With cancer diagnosis
* With diseases that require special dietary needs
* On urate-lowering medication within 3 months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Uric acid | 3 months
  Serum uric acid

SECONDARY OUTCOMES:
Body mass index | 3 months
  body mass index calculated from height and weight
Glucose metabolism | 3 months
  fasting glucose
Lipid profile | 3 months
  cholesterol
vitamin B12 | 3 months
  serum vitamin B12
holostranscobalamin | 3 months
  serum holotranscobalamin
homocysteine | 3 months
  serum homocysteine
vitamin D | 3 months
  serum 25(OH)D

CONTACTS AND LOCATIONS:
Overall Officials: Tina Hsueh-Ting Chiu, PhD, Principal Investigator — Fu-Jen Catholic University, Department of Nutritional Science
Locations (1):
- Department of Nutritional Science, Fu-Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared after the results have been published in peer review journals.